CLINICAL TRIAL: NCT05034016
Title: High Myopic Posterior Scleral Fixation System
Brief Title: The Exploratory Clinical Trials on the Primary Safety and Effectiveness of High Myopic Posterior Scleral Fixation System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: GuangZhou WeiShiBo Biotechnology Co., ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TREC2019-30.A2
Record Dates: First submitted 2021-08-26; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: High Myopia; Macular Schisis
Keywords: Posterior scleral reinforcement; Macular ischemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HM experimental group (Experimental): Intraocular implant test product
  Interventions: Device: High Myopic Posterior Scleral Fixation System
- Natural observation control group (No Intervention): Natural observation of the disease changes, no surgical intervention

INTERVENTIONS:
Device: High Myopic Posterior Scleral Fixation System — Implant HM into the eye through posterior scleral reinforcement
  Other Names: HM
  Arms: HM experimental group

SUMMARY:
The purpose of this study is to assess the primary safety and efficacy of High Myopic Posterior Scleral Fixation System in the treatment of macular schisis caused by high myopia.

DETAILED DESCRIPTION:
Posterior Scleral Reinforcement（PSR） is the only surgical method that can delay the the development of high myopia. However, The surgical method is restricted by the material source limitation and macular ischemia in the eye after reinforcement. The investigators have designed a new posterior scleral fixation system，Its basic material is medical silicone，The product is designed to solve the problem of material source limitation and macular ischemia in the eye after reinforcement.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~65, male or female;
2. Refractive ranges from -6.00d to -25.00d;
3. The axial length of the operative eye was 26-32mm;
4. Macular cleavage 200-1000μm;
5. Corrected visual acuity of the operative eye < 0.3;
6. Able to understand the purpose of the test, voluntarily participate and sign the informed consent form.

Exclusion Criteria:

1. Known allergy to silica gel and patients with scar constitution;
2. Ocular inflammation;
3. Fundus hemorrhage;
4. Macular hole;
5. Macular cleavage of the contralateral eye greater than 200μm;
6. Corrected visual acuity of contralateral eye < 0.4;
7. Opacity of the refractive medium;
8. Eye tumor;
9. History of hyperthyroidism;
10. Other ophthalmic concomitant diseases that cannot be controlled, such as diabetic retinopathy, hypertensive fundus lesions, optic nerve atrophy, etc.;
11. Severe impairment of liver and kidney function and/or severe systemic diseases (such as cardiovascular, respiratory, digestive, nervous, endocrine, genitourinary, etc., depending on the tolerance of surgery);
12. Women who are pregnant (determined by a blood pregnancy test at the first visit), who are preparing for pregnancy during the test, and who are breastfeeding;
13. a history of drug abuse or alcohol abuse;
14. participate in other drug or medical device clinical trials within 30 days prior to the screening of this clinical trial;
15. Any condition of the subject that the study physician considers to be an impediment to the clinical trial (e.g. subject's susceptibility to mental stress, uncontrollable mood, depression, etc.);
16. Poor compliance of the subject, unable to complete the test process as required.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-04-24 (Estimated)

PRIMARY OUTCOMES:
Macular reduction rate | 24 weeks
  24 weeks after implantation of the High Myopic Posterior Scleral Fixation System

SECONDARY OUTCOMES:
Best corrected visual acuity | Baseline (Before surgery), 1 day, 1 week, 4 weeks, 12 weeks, 24 weeks,
  ETDRS table
Axial length | Baseline (Before surgery), 24 weeks after surgery
  A-scan
Diopter | Baseline (Before surgery), 24 weeks after surgery
  Refractometer

CONTACTS AND LOCATIONS:
Overall Officials: Wenbing Wei, MD,Ph.D, Study Chair — Beijing Tongren Hospital
Locations (1):
- The First Affiliated Hospital of Guangzhou University of traditional Chinese Medicine, Guangzhou, Guangdong, China